CLINICAL TRIAL: NCT02246608
Title: Effect of Oasis® Wound Matrix on Stage III and IV Trunk Pressure Wounds Treated With Negative Pressure Wound Therapy (NPWT)
Brief Title: Effect of Oasis® Wound Matrix on Stage III and IV Trunk Pressure Wounds Treated With Negative Pressure Wound Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kettering Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHN-RSWound-P14-N01
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Open Wound Abdominal Wall; Wound Non Healing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine NPWT Standard of Care (Active Comparator): Prior to applying and activating the Negative Pressure Wound Treatment (NPWT) pump, standard of care dressing will be placed.
  Interventions: Device: Routine NPWT Standard of Care
- NPWT Standard of Care plus Oasis wound product (Experimental): Prior to applying and activating the Negative Pressure Wound Treatment (NPWT) pump, Oasis wound product will be applied in addition to standard of care dressing.
  Interventions: Device: NPWT Standard of Care plus Oasis wound product

INTERVENTIONS:
Device: NPWT Standard of Care plus Oasis wound product — Oasis® is a porcine acellular small intestine submucosa material compatible with human tissue. It is a complex scaffold that provides optimal environment for restoration of tissue structure. It guides tissue growth and traps growth factors. Oasis Matrix indications include partial and full thickness wounds and skin loss injuries as well as second-degree burns.
  Arms: NPWT Standard of Care plus Oasis wound product
Device: Routine NPWT Standard of Care — Specialized material, often foam, designed to protect the wound and promote healing during NPWT.
  Arms: Routine NPWT Standard of Care

SUMMARY:
This study evaluates the therapeutic effect of Oasis® Matrix along with Negative Pressure Wound Therapy (NPWT) on pressure wounds. Either Oasis or standard foam will be applied to the wound prior to activating the NPWT.

DETAILED DESCRIPTION:
In this study, patients being treated with Negative Pressure Wound Therapy (NPWT) will be randomized to receive either:

1. Oasis® matrix, applied to the wound, along with standard of care including NPWT OR
2. Standard foam, applied to the wound prior to activation of NPWT, which is standard care.

Wounds will be examined weekly for up to 12 weeks. At weeks 4, 8, and 12, the NPWT evacuation canister will be collected for specimen analysis.

The aim of this study is to determine the therapeutic effect of using Oasis® Wound Matrix with NPWT. Outcomes include: a) closure rate of non-healing wounds, and b) levels of growth factors and interleukins in fluid evacuated from the wound.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-89 who exhibit stage III or IV trunk pressure wounds with no signs of infection.
* HbA1C < 8 (if patient is diabetic)
* Adequate nutrition including albumin above 2.0 and prealbumin above 15.

Exclusion Criteria:

* Wounds that cannot have a NPWT device properly applied due to location (too close to anus), diarrhea, periwound skin issues.
* Patients with Infected wounds.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Simman, MD, Principal Investigator — Kettering Health Network
Locations (1):
- Kettering Medical Center, Kettering, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NPWT Standard of Care: Prior to applying and activating the Negative Pressure Wound Treatment (NPWT) pump, foam wound product will be applied.
  Routine NPWT plus foam wound product: Specialized material, often foam, designed to protect the wound and promote healing during NPWT.
- NPWT Standard of Care Plus Oasis Wound Product: Prior to applying and activating the Negative Pressure Wound Treatment (NPWT) pump, Oasis wound product will be applied.
  Routine NPWT plus Oasis wound product: Oasis® is a porcine acellular small intestine submucosa material compatible with human tissue. It is a complex scaffold that provides optimal environment for restoration of tissue structure. It guides tissue growth and traps growth factors. Oasis Matrix indications include partial and full thickness wounds and skin loss injuries as well as second-degree burns.
Period: Overall Study
Arm/Group | NPWT Standard of Care | NPWT Standard of Care Plus Oasis Wound Product
Started | 22 | 21
Completed | 10 | 11
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NPWT Standard of Care | NPWT Standard of Care Plus Oasis Wound Product | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Closure Rate of Non-healing Wounds
Description: Wound dimensions will be measured weekly and monitored for changes
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of healing
Arm/Group | NPWT Standard of Care | NPWT Standard of Care Plus Oasis Wound Product
Number analyzed (Participants) | 10 | 11
percentage of healing | 45.79 (38.72) | 89.98 (9.47)

2. Secondary Outcome: Growth Factors
Description: Fluid collected from the wound will be examined for the presence of growth factors and interleukins.
Time Frame: 12 weeks
Population: Data ended up not being collected for subjects and analysis was not completed for this outcome. Only have data on wound healing from wound measurements.
Arm/Group | NPWT Standard of Care | NPWT Standard of Care Plus Oasis Wound Product
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent to completion of 12 week study visit.
Description: The events and effects noted as documented Risks will not be reported unless the event carries a level of severity that is unexpected.
  Hospitalization due to subject co-morbidities unrelated to Wound Treatment in this at-risk population will not be considered an SAE.
Arm/Group | NPWT Standard of Care | NPWT Standard of Care Plus Oasis Wound Product
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/10 | 1/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPWT Standard of Care (N=10) | NPWT Standard of Care Plus Oasis Wound Product (N=11)
Gangrene (Vascular disorders) | 0 (0) | 1 (1)
Abdominal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Septic shock (Vascular disorders) | 1 (1) | 0 (0) — infection from PEG tube malfunction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT02246608/Prot_SAP_000.pdf